CLINICAL TRIAL: NCT05192824
Title: Effects of Different Designs of Orthokeratology Lens on Myopia Control and Visual Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Principal Investigator, Shuxian zhang, Director, Tianjin Eye Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TianjinEH-Orthokeratology lens
Record Dates: First submitted 2021-11-19; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Myopic Progression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single-vision glasses (No Intervention): Subjects wearing single-vision glasses CR-39
- Orthokeratology lenses group 1 (Experimental): Subjects wearing orthokeratology lenses of 5mm optical zone.
  Interventions: Device: Orthokeratology lens
- Orthokeratology lenses group 2 (Experimental): Subjects wearing orthokeratology lenses of 5.5mm optical zone.
  Interventions: Device: Orthokeratology lens
- Orthokeratology lenses group 3 (Experimental): Subjects wearing orthokeratology lenses of 6mm optical zone.
  Interventions: Device: Orthokeratology lens
- Orthokeratology lenses group 4 (Experimental): Subjects wearing orthokeratology lenses of 6mm optical zone and the increased height of peripheral reverse curve.
  Interventions: Device: Orthokeratology lens

INTERVENTIONS:
Device: Orthokeratology lens — The intervention was according to the design of different optical zone and peripheral reverse curve
  Other Names: Ortho-K
  Arms: Orthokeratology lenses group 1; Orthokeratology lenses group 2; Orthokeratology lenses group 3; Orthokeratology lenses group 4

SUMMARY:
This study was aimed to evaluate the effects of different Orthokeratology，including the size of central optical zone and the height of peripheral reverse curve, on myopia control and visual quality.

DETAILED DESCRIPTION:
This study was aimed to evaluate the effects of different Orthokeratology on myopia control and visual quality. The different optical zone of Orthokeratology lens was divided into 4 groups, ranged from 5.5 mm to 6 mm. And the control group subjects with the single glasses was included. The effectiveness of Orthokeratology was measured by axial length progression. The visual quality of subjects was evaluated by a questionnaire, contrast sensitivity and wavefront aberration.

ELIGIBILITY:
Inclusion Criteria:

* Myopia: between -1.00D and 4.00D in both eyes
* Astigmatism: <1.5D for with-the-rule astigmatism, <1.00D for the against-the-rule astigmatism
* Visual acuity: the best corrected vision acuity(BCVA)≥20/20 in both eyes
* Subjects that volunteer to participate in the clinical trial and sign informed consent

Exclusion Criteria:

* Contraindications of wearing Ortho-K.
* Diagnosis of strabismus, amblyopia and other refractive development of the eye or systemic diseases.
* Any type of strabismus or amblyopia
* Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
* Ocular conditions which might affect the refractive error (for example, cataract, ptosis)

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in axial length in 2 years | Every 6 months for a period 2 years
  The axial length was measured by AL-scan
Changes in Cycloplegic subjective refraction in 2 years | Every 6 months for a period 2 years
  The cycloplegic subjective refraction was evaluated by optometrist

SECONDARY OUTCOMES:
Change in visual questionnaire as compared to baseline（Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  The symptoms score measured by a visual questionnaire, each symptom was evaluated on a scale of 0 to 10.
Change in High-order aberrations (HOAs) in microns as compared to baseline(Postoperative 6 months, 12 months, 18 months and 24 months) | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  Ocular aberration measured by Zeiss i. Profiler Plus aberrometer
Change in contrast sensitivity as compared to baseline(Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  Contrast sensitivity measured by Stereo optical 6500
Change in choroidal thickness captured by Optical Coherent Tomographer (OCT) as compared to baseline(Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  choroidal thickness captured by Optical Coherent Tomographer (OCT) and measured using a customized software
Change in Corneal epithelial thickness captured by Optical Coherent Tomographer (OCT) as compared to baseline(Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  Corneal epithelial thickness captured by Optical Coherent Tomographer (OCT) customized software
Change in corneal biomechanics parameters (SSI) as compared to baseline (Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  Corneal response parameters(SSI) was evaluated by Corvis ST.
Change in peripheral refraction as compared to baseline (Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  Peripheral refraction measured by multispectral refraction topography
Change in corneal surface regularity index (SRI) as compared to baseline (Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  The corneal surface regularity index (SRI) was measured by Corneal Topography.
Change in corneal surface asymmetry index (SAI) as compared to baseline (Postoperative 6 months, 12 months, 18 months and 24 months） | baseline, postoperative 6 months, 12 months, 18 months and 24 months
  The corneal surface asymmetry index (SAI) was measured by Corneal Topography.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He M, Du Y, Liu Q, Ren C, Liu J, Wang Q, Li L, Yu J. Effects of orthokeratology on the progression of low to moderate myopia in Chinese children. BMC Ophthalmol. 2016 Jul 27;16:126. doi: 10.1186/s12886-016-0302-5. PMID 27464993
- [Background] Huang J, Wen D, Wang Q, McAlinden C, Flitcroft I, Chen H, Saw SM, Chen H, Bao F, Zhao Y, Hu L, Li X, Gao R, Lu W, Du Y, Jinag Z, Yu A, Lian H, Jiang Q, Yu Y, Qu J. Efficacy Comparison of 16 Interventions for Myopia Control in Children: A Network Meta-analysis. Ophthalmology. 2016 Apr;123(4):697-708. doi: 10.1016/j.ophtha.2015.11.010. Epub 2016 Jan 27. PMID 26826749
- [Background] Hu Y, Wen C, Li Z, Zhao W, Ding X, Yang X. Areal summed corneal power shift is an important determinant for axial length elongation in myopic children treated with overnight orthokeratology. Br J Ophthalmol. 2019 Nov;103(11):1571-1575. doi: 10.1136/bjophthalmol-2018-312933. Epub 2019 Jan 31. PMID 30705043
- [Background] Paune J, Fonts S, Rodriguez L, Queiros A. The Role of Back Optic Zone Diameter in Myopia Control with Orthokeratology Lenses. J Clin Med. 2021 Jan 18;10(2):336. doi: 10.3390/jcm10020336. PMID 33477514
- [Background] Gifford P, Tran M, Priestley C, Maseedupally V, Kang P. Reducing treatment zone diameter in orthokeratology and its effect on peripheral ocular refraction. Cont Lens Anterior Eye. 2020 Feb;43(1):54-59. doi: 10.1016/j.clae.2019.11.006. Epub 2019 Nov 24. PMID 31776061